CLINICAL TRIAL: NCT00523081
Title: Brief, Primary Care Cognitive Behavioral Therapy (CBT) for Unmedicated Youth
Brief Title: Study of Adolescence and Depression
Acronym: STAND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH073918-01A1 (NIH); R01MH073918-01A1 (NIH)
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2012-07

CONDITIONS: Major Depressive Disorder
Keywords: adolescent depression treatment, cognitive behavioral therapy,; collaborative care
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Teens in the experimental group will meet with a research counselor for five to nine individual, 50-minute weekly sessions. They will learn ways to deal with stress and feel better. The study counselor will also talk to the teen's doctor from time to time to help plan for the best possible care.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Active Control (Active Comparator)
  Interventions: Behavioral: Active control

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy (CBT) — Half the teens in the study will also meet with a research counselor for five to nine individual, weekly sessions that last about 50 minutes each. Whether a teen attends the weekly counseling sessions is decided by chance, like flipping a coin. If teens are assigned to these sessions, they will learn ways to deal with stress and feel better. If teens take part in the counseling sessions, the study counselor will also talk to the teen's doctor from time to time to help plan for the best possible care.
  Arms: Experimental
Behavioral: Active control — Teens in the active control arm will keep seeing their doctor as usual. Teens and a parent are interviewed briefly over the phone to see if they are appropriate for the study. If they qualify for the study, there is an hour-long interview with teen over the telephone and a 30 minute interview with the parent. They will be interviewed six more times in the next two years.
  Arms: Active Control

SUMMARY:
STAND is a research study testing a way to help teens between 12-18 years of age who have symptoms of sadness or depression. The study hopes to learn if teens do better if they get five to nine counseling sessions of cognitive behavioral therapy coordinated with the support of their doctor. All teens who join the study will keep seeing their doctor as usual.

Teens and a parent are interviewed briefly over the phone to see if they are appropriate for the study. If they qualify for the study, there is an hour-long interview with teen over the telephone and a 30 minute interview with the parent. The interview will include questions about the teen's mood, feelings, behavior, and how they get along with friends and family members. The parent is also asked about his or her own feelings and mood. If the teen and parent join the study, they will be interviewed six more times in the next two years.

Half the teens in the study will also meet with a research counselor for five to nine individual, weekly sessions that last about 50 minutes each. Whether a teen attends the weekly counseling sessions is decided by chance, like flipping a coin. If teens are assigned to these sessions, they will learn ways to deal with stress and feel better. If teens take part in the counseling sessions, the study counselor will also talk to the teen's doctor from time to time to help plan for the best possible care.

DETAILED DESCRIPTION:
Substantial numbers of depressed adolescents either decline antidepressant medication or quickly discontinue such medications before benefits are expected. Recent controversies regarding the safety of SSRI anti-depressants are likely to increase medication refusal. More than half of depressed adolescents identified in primary care prefer psychosocial treatments, compared to 20% who prefer medication. Among the psychotherapy alternatives to medication, cognitive behavioral therapy (CBT) has the strongest research support.

The STAND study is a two-arm, randomized, efficacy-effectiveness trial in primarily a Health Maintenance Organization (HMO), comparing a treatment as usual (TAU) control condition to TAU plus brief, individual, collaborative care CBT delivered in primary care. We will enroll 240 youth ages 12 to 18 who, during this depressive episode, have either declined anti-depressant medication or who received a single dispense of anti-depressant medication but quickly discontinued. All enrolled cases will be reassessed periodically throughout a 24-month follow-up period. The primary clinical outcome is recovery from the index episode of major depression, assessed via research diagnosis. Secondary outcomes include continuous depression symptomatology; depression response; rates of new, recurrent episodes of major depression in the follow-up period; improvements in psychosocial function; clinical improvement; reduction in depression-related dysfunction; parent/youth attitudes regarding treatment. We will also examine incremental cost-effectiveness of CBT compared to TAU from the HMO, family, and societal perspectives. We will conduct exploratory analyses of mediation and moderation of depression treatment outcomes, and employ data from the TAU control condition to estimate the usual outcomes for depressed youth who refuse/discontinue antidepressant medication. Finally, we will examine how provider, parent and youth barriers, attitudes and beliefs moderate outcomes, as well as possibly change over time as a function of participation in this program.

The validation of a primary care model for brief CBT may prove to be a significant benefit to the sizeable numbers of depressed youth identified in primary care, and who elect not to try anti-depressant medication or quickly discontinue an initial trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-18
* Current diagnosis of Major Depressive Disorder

Exclusion Criteria:

* Psychosis
* Bipolar
* Taking anti-depressant medication
* Significant intellectual impairment
* Recent treatment with cognitive behavioral therapy

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 212 (Actual)
Dates: Start 2006-10; Primary Completion 2012-03 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The two Primary outcomes are (a) recovery of response from the index episode of major depression and (b) improvements in continuous depression symptomatology . | Assessment at 1 3, 6,12, 18 and 24 months,

SECONDARY OUTCOMES:
Secondary outcomes include depression response; rates of new, recurrent episodes of MDD during follow-up; improvement in psychosocial function; clinical improvements; and reduction in depression-related dysfunction. | Assessment at 1 3, 6,12, 18 and 24 months,

CONTACTS AND LOCATIONS:
Overall Officials: Greg N Clarke, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States

REFERENCES:
- [Derived] Dickerson JF, Lynch FL, Leo MC, DeBar LL, Pearson J, Clarke GN. Cost-effectiveness of Cognitive Behavioral Therapy for Depressed Youth Declining Antidepressants. Pediatrics. 2018 Feb;141(2):e20171969. doi: 10.1542/peds.2017-1969. Epub 2018 Jan 19. PMID 29351965